CLINICAL TRIAL: NCT06951373
Title: Comparison of Pain, Cosmesis and Early Restoration of Breast Feeding in Multiple Percutaneous Needle Aspiration Vs Incision and Drainage for Small Breast Abscess Management
Brief Title: Comparison of Multiple Percutaneous Needle Aspiration Versus Incision and Drainage in Small Breast Abscesses: Pain, Cosmesis, and Early Breastfeeding Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Quaid-e-Azam Medical College (Other)
Responsible Party: Principal Investigator, Aroona Arif, Postgraduate Resident, Quaid-e-Azam Medical College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: No. PG656/DME/QAMC/BWP
Record Dates: First submitted 2025-03-20; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Breast Abscess
MeSH Terms: interventions — Drainage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Multiple Percutaneous Needle Aspiration (MPNA) Group (Experimental): Participants in this group underwent multiple percutaneous needle aspiration for the treatment of small breast abscesses
  Interventions: Procedure: Multiple Percutaneous Needle Aspiration (MPNA); Procedure: Incision and Drainage (ID)
- Incision and Drainage (ID) Group (Active Comparator): Participants in this group underwent incision and drainage for the treatment of small breast abscesses.
  Interventions: Procedure: Multiple Percutaneous Needle Aspiration (MPNA); Procedure: Incision and Drainage (ID)

INTERVENTIONS:
Procedure: Multiple Percutaneous Needle Aspiration (MPNA) — A minimally invasive technique involving repeated needle aspiration of breast abscess fluid without making an incision.
Procedure: Incision and Drainage (ID) — A surgical procedure involving an incision in the abscess to allow drainage of pus, followed by wound care.

SUMMARY:
This study aims to compare the effectiveness of multiple percutaneous needle aspiration (MPNA) versus incision and drainage (ID) for the management of small breast abscesses in breastfeeding women. The trial evaluates three key outcomes: post-procedure pain levels, cosmetic satisfaction, and the timing of breastfeeding restoration. The study is conducted at the Department of Surgery, Bahawal Victoria Hospital Bahawalpur, enrolling 110 lactating women aged 18-45 years with abscesses ≤5 cm in diameter. Participants were treated with either MPNA or ID based on clinical decision and patient preference. Pain levels were assessed using a standardized scale, cosmetic outcomes were evaluated via patient-reported satisfaction, and breastfeeding restoration was monitored at baseline, one week, and one month post-treatment. Findings indicate that MPNA is associated with lower pain scores, better cosmetic satisfaction, and faster resumption of breastfeeding compared to ID, suggesting MPNA as a preferred first-line treatment for small breast abscesses.

ELIGIBILITY:
Inclusion Criteria:

* Married breastfeeding women Age: 18-45 years Diagnosed with breast abscess (≤5 cm in diameter)

Exclusion Criteria:

* Complicated abscesses Compromised immune system History of prior surgical interventions for breast abscess Unwilling to participate in the study

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 110 (Actual)
Dates: Start 2021-01-09 (Actual); Primary Completion 2021-06-08 (Actual); Study Completion 2021-06-08 (Actual)

PRIMARY OUTCOMES:
Pain Score | 1 week post-procedure
  Assessment of pain using a standardized visual analog scale (VAS) at 1 week after the procedure.
Breastfeeding Restoration | 1 month post-procedure
  Proportion of patients resuming breastfeeding at 1 month after intervention, determined by patient self-report.

SECONDARY OUTCOMES:
Cosmetic Satisfaction | 1 month post-procedure
  Patient-reported satisfaction with cosmetic outcomes, assessed through a survey at 1 month after intervention.

CONTACTS AND LOCATIONS:
Locations (1):
- Bahawal Victoria Hospital, Bahawalpur, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No